CLINICAL TRIAL: NCT06893068
Title: Evaluation of a Multimodal Model-Based Clinical Intelligent Management System: A Pragmatic Randomized Controlled Trial
Brief Title: Clinical Intelligent Management System Pragmatic RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tsinghua University (Other)
Responsible Party: Principal Investigator, Tien Yin Wong, Professor, Tsinghua University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-22
Record Dates: First submitted 2025-02-12; First posted 2025-03-25 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Primary Care Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assist group (Experimental): Physicians in the intervention group will employ the intelligent management system with AR glasses to assist in diagnosis and treatment, while patients will interact with the system's patient interface to access health education, follow-up reminders, and AI-powered home consultation features.
  Interventions: Device: AI-based clinical intelligent management system
- Traditional group (No Intervention): Physicians in the control group will conduct routine diagnoses and treatments, while patients will receive standard health education and follow-up care.

INTERVENTIONS:
Device: AI-based clinical intelligent management system — The clinical intelligent management system, integrated with AR glasses and powered by a multimodal foundational model, is designed to improve the quality of outpatient care at community health service centers.
  Arms: AI-assist group

SUMMARY:
This study aims to evaluate the effectiveness of a clinical intelligent management system, based on a multimodal foundational model, in improving the quality of primary care at a community health service center.

Using a prospective, randomized controlled, single-blind study design, the trial will include primary care physicians and adult patients seeking care at the Tiantongyuanbei Community Health Service Center and Shanghai Health and Medical Center.

Physicians in the intervention group will utilize the intelligent management system with AR glasses to aid in diagnosis and treatment, while patients will engage with the system's patient interface to access health education, follow-up reminders, and AI-powered home consultation features. In contrast, physicians in the control group will provide routine diagnoses and treatments, with their patients receiving standard health education and follow-up care. The trial was designed with the assistance of a digital twin-based clinical research system (termed X Town).

By comprehensively evaluating diagnostic quality, physicians' clinical abilities, patient-reported outcomes, and system appraisals, this study will assess the effectiveness of the clinical intelligent management system in enhancing the quality of primary care and patient management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Receiving care at a community health service center
* Able to understand and comply with the study procedures
* Agrees to participate in the study and signs the informed consent form

Exclusion Criteria:

* Patients with severe mental illness
* Patients unable to independently complete the questionnaire
* Patients expected to be unable to complete follow-ups within three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-04-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Assessment of clinical performance | From enrollment to the end of treatment at 3 months of all recruited cases
  Primary Care Quaility Assessment Scales (range: 0 to 100 for each case; the higher scores means the better performance)

SECONDARY OUTCOMES:
AI-System's appraisal | At the end of 3 months
  System usability was accessed by participating doctors of an AI-assisted group using the Health Information Technology Usability Evaluation Scale, rated on a five-point Likert scale from strongly disagree (1) to strongly agree (5). (A higher scale value indicates higher perceived usability of the technology.)

CONTACTS AND LOCATIONS:
Overall Officials: Tien Yin Wong, Principal Investigator — Tsinghua University
Locations (1):
- Shanghai Health and Medical Center, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No